CLINICAL TRIAL: NCT01347203
Title: A Randomized, Open-label, 4-period Crossover Study to Evaluate the Pharmacokinetics (PK), Pharmacodynamics (PD) and the PK/PD Relationship of DPOC-4088 After Single Oral Dosing of 100 and 200 mg in 2 Prolonged Release Formulations (16 and 20 hr) in 12 Healthy Young Male Subjects
Brief Title: A Healthy Volunteer Study to Evaluate for a Single Dose of 4 Different Tablets of DPOC-4088 the Absorption and Elimination From the Body and the Potential Effect on Blood Clotting
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Diakron Pharmaceuticals (Industry)
Responsible Party: Stephane E. Allard, Diakron Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DPOC-001
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Deep Vein Thrombosis Leg
Keywords: phase I; healthy volunteers; crossover study; pharmacokinetics; pharmacodynamics
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): DPOC-4088 prolonged release tablet 100 mg (Formulation A= 16 hr release formulation)
  Interventions: Drug: DPOC-4088
- Treatment B (Experimental): DPOC-4088 prolonged release tablet 200 mg (Formulation A= 16 hr release formulation)
  Interventions: Drug: DPOC-4088
- Treatment C (Experimental): DPOC-4088 prolonged release tablet 100 mg (Formulation B= 20 hr release formulation)
  Interventions: Drug: DPOC-4088
- Treatment D (Experimental): DPOC-4088 prolonged release tablet 200 mg (Formulation B= 20 hr release formulation)
  Interventions: Drug: DPOC-4088

INTERVENTIONS:
Drug: DPOC-4088 — A single oral dose of DPOC-4088 prolonged release tablet 100 mg (Formulation A = 16 hr release formulation)
  Arms: Treatment A
Drug: DPOC-4088 — A single oral dose of DPOC-4088 prolonged release tablet 200 mg (Formulation A = 16 hr release formulation)
  Arms: Treatment B
Drug: DPOC-4088 — A single oral dose of DPOC-4088 prolonged release tablet 100 mg (Formulation B = 20 hr release formulation)
  Arms: Treatment C
Drug: DPOC-4088 — A single oral dose of DPOC-4088 prolonged release tablet 200 mg (Formulation B = 20 hr release formulation)
  Arms: Treatment D

SUMMARY:
This will be a study existing of 4 periods, to evaluate for a single dose of 4 different tablets of DPOC-4088 the absorption and elimination from the body and the potential effect on blood clotting. The differences between the tablets are the dose (100 or 200 mg) and the rate of release of DPOC-4088 from the tablet (16 or 20 hours). The allocation of the tablets in each period will be determined by chance but is known upfront.

DETAILED DESCRIPTION:
This will be a randomized, open-label, single oral dose study. The 4-period crossover study will determine and compare the PK and PD profiles of DPOC-4088 when administered as a single oral dose of 100 mg and 200 mg of DPOC-4088 in two prolonged release formulations (16 and 20 hr) in 12 evaluable young healthy male subjects.

Each subject (in a fasting state) will receive each of the 4 treatments (A, B, C, and D) in a balanced, 4-period crossover design. Each treatment consists of a single oral dose of 100 mg or 200 mg of DPOC-4088 in either prolonged release formulation (16 or 20 hr). Subjects will arrive at the study unit for an overnight fast of at least 10 hrs the evening before each dosing period and remain in the unit for at least 24 hrs after dosing. Standard meals will be provided and subjects will receive their first meal after dosing at 4 hrs post-dose. Blood samples will be drawn for PK and PD evaluations immediately prior to dosing and at specified time intervals for 48 hrs post-dosing. Each dosing period will be separated by at least a 5-day washout period that is preferentially not to exceed 10 days.

In healthy young male subjects, the safety, tolerability, and the PK profile of DPOC-4088 will be assessed. Additionally, this study will assess the PD profile and the relationship of PK/PD in terms of the ability of DPOC-4088 to inhibit thrombin activity (based on prolongation of aPTT, ECT, TT and PT).

ELIGIBILITY:
Inclusion Criteria:

1. Male between 18 to 45 years of age.
2. Either a non- or a light-smoker (<5 cigarettes per day) and agrees to refrain from smoking during the entire 4-week study until after the last PK sample is drawn.
3. Body-mass index (BMI) of 18-30 kg/m2.
4. In good health on the basis of history, physical examination, and routine laboratory data.
5. Understands the procedures and agrees to participate in the study program by giving written informed consent.
6. Coagulation tests including aPTT, ECT, TT and PT within the reference range and a platelet count >145,000/mm3.
7. At screening, normal transaminases and negative Hemoccult Sensa test. In the event of a positive Hemoccult test, the test should be repeated twice. If the results of both repeats tests are negative, the first Hemoccult test result is considered a false positive and the subject may be included.

Exclusion Criteria:

1. Mentally or legally incapacitated, significant emotional problems at the time of the study, or a history of psychiatric disorders.
2. History within the last 10 years of asthma or other pulmonary disease, major cardiovascular, hepatic, endocrine (including diabetes), rheumatological, or renal disease or of prior spine or disc surgery.
3. History within the last 10 years of neurologic disease including stroke, transient ischemic attacks, seizure, head trauma, neurological tumors, brain or spinal cord surgery, neuropathy, or neuromuscular illness.
4. Active gastrointestinal disease including: peptic ulcer disease, gastritis, clinically significant Helicobacter pylori infection, inflammatory bowel disease, diverticular disease, colonic polyps, or of any gastrointestinal malignancy, or recent (within 3 weeks) benign enteritis.
5. History of any illness or condition that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering study drug to the subject (e.g., surgery within the previous 3 months).
6. Donated a unit of blood (450 mL) or participated in another clinical study drug trial within the 4 weeks prior to screening.
7. Family or personal history of bleeding disorders, including von Willebrand's disease.
8. History of significant gingivitis or other periodontal disease.
9. Received any prescription anticoagulant within the 30 days preceding screening including but not limited to warfarin, heparin, low-molecular weight heparin, hirulog, hirudin, argatroban, or dabigatran.
10. Has received 14 days prior to first dosing or anticipates needing during the study any prescription or nonprescription (including over the counter) preparation that contains aspirin (including low-dose aspirin), ibuprofen, indomethacin, diclofenac, naproxen, meloxicam, any other NSAID or NSAID-containing product such as pain relievers, cold or sinus remedies, or any other drug which influences platelet aggregation.
11. Received any investigational drug within the 30 days preceding screening.
12. Regular user of any medication (including over-the-counter medication) for 14 days prior to first dosing, except for acetaminophen. Subject currently uses prescription or nonprescription drugs on a regular basis which cannot be discontinued for 14 days prior to first dosing until the last study visit (including "recreational use" of illicit drugs). Subject has a recent history (within the last 2 years) of drug or alcohol abuse.
13. Subjects unable to stop using the following medications during the study (from first dosing until after the last study visit): erythromycin or erythromycin-like drugs, clarithromycin, diltiazem, cimetidine, warfarin-like anticoagulants, cyclosporine, itraconazole (or other systemic antifungal agents in the azole class), nefazodone, selective serotonin reuptake inhibitors (SSRI antidepressants), benzodiazepines, any systemic immunosuppressive agents (including glucocorticoids), cisapride and the H1 antagonists terfenadine and astemizole, and HIV protease inhibitors.
14. Unable to refrain from the use of antacids, H2 blockers, sucralfate, or proton pump inhibitors beginning 14 days prior to first dosing until the last study visit.
15. Has had minor or major surgery (including dental surgery) within previous 3 months prior to first dosing or is anticipated to have minor or major surgery (including dental surgery) within 2 weeks after completion of the study.
16. Positive hepatitis serology (HBsAg and anti-HCV) showing any sign of active hepatitis.
17. History of any chronic and/or active hepatic disease including hepatitis or biliary tract disease. Any subject with a history of hepatitis B or C at screening will be excluded. Subjects with a history of self-limited hepatitis A with complete resolutions documented at ≥12 months prior to entry would be eligible for inclusion.
18. Significant unexplained and/or reproducible abnormalities on prestudy clinical examination or laboratory measurements.
19. History of significant drug allergy or any clinically significant adverse event of a serious nature related to the administration of either a marketed or investigational drug.
20. Known history of fainting from phlebotomy or from minor trauma resulting in bleeding.
21. Habitual heavy consumer of coffee (more than 6 cups of coffee/day).
22. Unable to refrain from consumption of grapefruit or grapefruit juice for at least 14 days prior to first dosing until the last study visit.
23. Unable to refrain from the use of St. Johns wort for at least 14 days prior to first dosing until the last study visit.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
plasma concentration ratios | pre-dose until 48 hrs post-dose
  Cmax/C12 hr and Cmax/C24 hr for each of the 2 doses and 2 prolonged release formulations of DPOC-4088

SECONDARY OUTCOMES:
other pharmacokinetics | pre-dose until 48 hrs post-dose
  AUC 0-48 hr, AUC0-∞, Cmax, C12 hr, C24 hr, Tmax, T1/2
blood coagulation | pre-dose until 48 hrs post-dose
  aPTT, ECT, TT and PT
safety | throughout clinical trial
  adverse events and abnormal laboratory findings

CONTACTS AND LOCATIONS:
Overall Officials: Luc M Van Bortel, Prof. dr., Principal Investigator — University Ghent
Locations (1):
- Drug Reseach Unit Ghent, Ghent, Belgium